CLINICAL TRIAL: NCT00004662
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Dehydroepiandrosterone in Women With Active Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11918; NU-584
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: arthritis & connective tissue diseases; immunologic disorders and infectious disorders; rare disease; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Connective Tissue Diseases; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: dehydroepiandrosterone

SUMMARY:
OBJECTIVES:

I. Evaluate the safety and efficacy of synthetic dehydroepiandrosterone, GL701, in women with active systemic lupus erythematosus.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are stratified by participating institution.

Patients are randomly assigned to daily oral dehydroepiandrosterone or placebo for 52 weeks. Patients are evaluated every 13 weeks on study and return for a follow-up 6 weeks after completion of therapy.

Concurrent therapy with estrogen replacement and stable doses of prednisone, azathioprine, methotrexate (with folate supplementation), hydroxychloroquine, and nonsteroidal anti-inflammatory drugs is allowed. Other investigational medications and immunosuppressants are prohibited.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Systemic lupus erythematosus by 1982 American College of Rheumatology criteria Diagnosed for at least 6 months

Systemic Lupus Activity Measure score at least 7 Points for erythrocyte sedimentation rate excluded

SLEDAI score of greater than 2 at both screening and qualifying visits

--Prior/Concurrent Therapy--

No prior participation in any dehydroepiandrosterone (DHEA) study

No investigational agent within the longer of 30 days or 10 half-lives of the agent

Prednisone (or equivalent) dose 0 to 10 mg/day Unchanged for at least 6 weeks prior to entry

At least 3 months since immunosuppressants other than azathioprine and methotrexate, including:

* DHEA
* Adrenocorticotropin hormone
* Androgens
* Cyclophosphamide
* Cyclosporine
* Immune globulin

At least 6 weeks since change in azathioprine, methotrexate, or hydroxychloroquine

--Patient Characteristics-- Renal: No requirement for hemodialysis

Cardiovascular: No serious abnormality on electrocardiogram

Other:

* No hypersensitivity to DHEA or inactive ingredients in GL701 formulation, i.e., cornstarch, lactose, or magnesium stearate
* No history of breast cancer or reproductive tract malignancy
* Cervical carcinoma eligible if surgically cured, i.e., no evidence of disease for 5 years
* No condition that would prevent compliance or follow-up, e.g.: Alcoholism Drug addiction Acute withdrawal from chemical dependency
* Psychiatric disease
* No pregnant or nursing women
* Negative pregnancy test required of fertile women
* Reliable contraception required of fertile women
* No estrogen-containing oral contraceptives on study
* At least 3 weeks since estrogen-containing oral contraceptives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1996-03

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Ramsey-Goldman, Study Chair — Northwestern University